CLINICAL TRIAL: NCT06720623
Title: Diagnostic Power of Basal LH Compared to Peak LH After Stimulus Test in the Diagnosis of Central Precocious Puberty
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LuteoTest
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Central Precocious Puberty (CPP)
Keywords: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational, retrospective, single-center study focused on the diagnosis of Central Precocious Puberty in female patients.

DETAILED DESCRIPTION:
The study enrolls female patients undergoing GnRh testing for suspected diagnosis of Central Early Puberty between january 2017 and December 2020 at the Pediatrics Unit of IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola.

The study design provides 2 cohorts of female patients on the basis of the LH peak value in GnRH test: patients with LH peak value < 5U/L, and patients with LH peak value > 5U/L.

The primary aim is to assess the diagnostic power of basal LH comparing with the LH peak value after stimulus test with GnRH in female patients with suspected precocious puberty. The secondary aim is to assess the association of the following variables between the two cohorts: uterine volume, longitudinal uterine diameter, presence of endometrial rhyme, ratio of peak LH/FSH values and dose per kg of GnRH administered during stimulus test.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with onset of signs of early pubertal development (onset of telarche) before the age of 8 years, who referred to the Pediatrics Unit of IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola between January 2017 and December 2020;
* Female patients undergoing GnRh testing for suspected diagnosis of Central Early Puberty between january 2017 and December 2020;
* Obtaining informed consent from parents/legal guardian of pediatric patients.

Exclusion Criteria:

• Patients with Peripheral precocious puberty.

Max Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Female patients undergoing GnRh testing for suspected diagnosis of Central Early Puberty between january 2017 and December 2020 at the Pediatrics Unit of IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
LH value | at baseline
  basal Lh value, and LH peak value after stimulus test with GnRH (mU/mL )

SECONDARY OUTCOMES:
Uterine volume | at baseline
  ml
Longitudinal uterine diameter | at baseline
  mm
Presence of endometrial rhyme | at baseline
  yes/no
Ratio of peak LH/FSH values | at baseline
  peak LH (mU/mL) value / FSH value ( mU/mL)
peak LH (mU/mL) value / FSH value ( mU/mL) | at baseline
  mcg/kg

CONTACTS AND LOCATIONS:
Overall Officials: Federico Baronio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

REFERENCES:
- See also: PubMed article "Does Basal Morning Luteinizing Hormone (bLH) Predict Central Precocious Puberty (CPP) in Girls?" — https://pubmed.ncbi.nlm.nih.gov/38541222/